CLINICAL TRIAL: NCT03602651
Title: MAGZEN® Effect on Recent Anxiety Reaction (STRESS2)
Brief Title: MAGZEN® Effect on Recent Anxiety Reaction
Acronym: STRESS2
Status: Completed | Type: Observational
Sponsor: Laboratoire Dielen (Industry)
Responsible Party: Sponsor
Other Study IDs: N°ID-RCB : 2018-A01516-49
Record Dates: First submitted 2018-07-18; First posted 2018-07-27 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MAGZEN®: All patient will be treated with MAGZEN® and will be evaluated with the Hamilton-anxiety scale (HAM-A)
  Interventions: Other: Hamilton-anxiety scale (HAM-A)

INTERVENTIONS:
Other: Hamilton-anxiety scale (HAM-A) — Evolution of anxiety disorders is evaluated by the Hamilton-anxiety scale (HAM-A)

SUMMARY:
Multicentres, observational study, prospective, to evaluate the effect of MAGZEN® in the treatment of recent anxiety reaction.

DETAILED DESCRIPTION:
107 patients suffering from recent anxiety reaction will be included in the study. They will be treated by MAGZEN® during 4 weeks and we will study the effect of this treatment on the evolution of their anxiety after the cure.

ELIGIBILITY:
Inclusion Criteria:

* patient suffering from recent anxiety reaction
* Hamilton-anxiety score ≥ 20 at inclusion
* recent anxiety disorders (less than 3 months) not treated by pharmacological or psychological treatment

Exclusion Criteria:

* major depressive syndrome
* anxiety disorders more than 3 months
* anxiety due to death

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients suffuring from a recent anxiety reaction not already treated.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
number of "responders patients" | 4 weeks
  number (%) of "responders patients" with a diminution of the HAM-A score ≥ 50 %

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric MD ROUILLON, Study Chair — Hôpital St Anne
Locations (1):
- Private practice, Marseille, France

IPD SHARING:
Plan to Share IPD: No